CLINICAL TRIAL: NCT03906773
Title: Validation of a Novel EHR Patient Portal Advance Care Planning Delivery System
Brief Title: Advance Care Planning GuideTailored for Primary Care Patients
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Seuli Brill, Associate Professor of Clinical Medicine, Ohio State University
Other Study IDs: 2015H0350
Record Dates: First submitted 2018-02-26; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Advance Care Planning; Chronic Disease; Communication Research
MeSH Terms: conditions — Chronic Disease | interventions — Advance Care Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The investigators seek to conduct a pragmatic trial including 2 sister clinical sites to test an innovation using a patient portal framework for Advance Care Planning. The intervention site implemented the intervention (secure patient portal delivered pre-visit planning framework for Advance Care Planning communication). The presence of ACP and the quality of documentation will be assessed through post-intervention chart review. Practice level enrollment was sought for the trial, and the framework will be delivered to all patients during a period of roll out. About 250 patients will receive the intervention.
  Interventions: Other: Patient Centered Medical Home Based Electronic Framework for Advance Care Planning
- control: The control site delivered usual care during the same period of roll out.

INTERVENTIONS:
Other: Patient Centered Medical Home Based Electronic Framework for Advance Care Planning — The intervention tested a pre-visit ACP workflow centered around a framework sent via secure Electronic Health Record (EHR)-linked patient portal in a real world clinical setting. The primary objectives were to determine its impact on frequency and quality of ACP documentation.
  Other Names: Secure patient portal delivered pre-visit planning for advance care planning
  Groups: Intervention

SUMMARY:
this project seeks to: validate results of ACP framework pilot study in a larger randomized controlled trial (rates and quality of ACP documentation) prior to using participatory design to develop an Electronic Health Record (EHR)-tethered patient portal delivered ACP communication guide, tailored for use in busy primary care settings, incorporating patients, caregivers, and primary care providers

ELIGIBILITY:
Inclusion Criteria:

* must have an activated patient portal account over 50 years of age scheduled for a well visit appointment or chronic visit follow up English speaking

Exclusion Criteria:

* under 50
* inactive patient portal account

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators seek to test participant intervention in a pragmatic primary care environment to the patient populations described above.
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Presence of Advance Care Planning (ACP) documentation as noted in description | 4 weeks post-intervention
  Presence of Electronic Health Record problem list based ACP documentation or presence of Electronic Health Record scanned completed Advance Directive document

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No